CLINICAL TRIAL: NCT07242768
Title: Regular Physical Exercise in Patients With Symptomatic Intracranial Arterial Stenosis: Three-year Follow-up of RESIST Trial
Brief Title: Follow-up Extension Study of Regular Physical Exercise in Patients With Symptomatic Intracranial Arterial Stenosis
Acronym: RESIST-FE
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor of Neurology, Xuanwu Hospital, Capital Medical University, Capital Medical University
Other Study IDs: SPORTS1102
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: Ischemic Stroke; Transient Ischemic Attack; Symptomatic intracranial arterial stenosis
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regular Physical Exercise Group: Participants with symptomatic ICAS who were assigned to the regular physical exercise intervention in the RESIST trial and completed the 12-month follow-up.
  Interventions: Other: Non-Interventional Study
- Control Group: Participants with symptomatic ICAS who were assigned to the control group in the RESIST trial and completed the 12-month follow-up.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — After completing 12-month intervention from RESIST trial, investigators would not make any interventions or impact on subjects.

SUMMARY:
This study will include the subjects with symptomatic intracranial arterial stenosis (ICAS) who have participated in and completed the 1-year follow-up of RESIST trial (NCT06615726). The aim is to observe the long-term clinical outcomes over 3 years after a 1-year regular physical exercise intervention in patients with symptomatic ICAS.

DETAILED DESCRIPTION:
This is a non-interventional, observational study designed to investigate long-term clinical outcomes in symptomatic ICAS patients who have already enrolled in RESIST trial and completed the 1-year follow-up.

After completing 12-month randomized intervention from RESISR trial, investigators continue to follow the subjects up to 3 years without any further intervention or changes to routine clinical management. The primary endpoint is the incidence of new ischemic stroke within 3 years. Secondary endpoints include new ischemic stroke and transient ischemic attack events in the responsible vessel supply area within 3 years; new ischemic stroke and transient ischemic attack events within 3 years; hemorrhagic stroke event within 3 years; myocardial infarction within 3 years; falls within 3 years; all-cause death within 3 years; the proportion of patients with modified Rankin Scale score 0-1 at 3 years; the score of mini-Montreal Cognitive Assessment at 3 years; and the score of EuroQol 5-Dimension 5-Level at 3 years.

Approximately 1,300 subjects who have completed the RESIST trial's 1-year follow-up and consented to continue will be included. The overall study duration will extend from the first participant's entry into the observation period until the last participant completes the 3-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who enrolled in the RESIST trial and completed the 12-month follow-up.
2. Written informed consent to participate in this 3-year observational extension.

Exclusion Criteria:

Participants who withdrew consent in the RESIST trial, decline to participate in this extension, or were lost to follow-up at 12 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include the subjects who enrolled in the RESIST trial.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
New ischemic stroke events | Within 3 years after randomization

SECONDARY OUTCOMES:
New ischemic stroke and transient ischemic attack events in the responsible vessel supply area | Within 3 years after randomization
New ischemic stroke and transient ischemic attack events | Within 3 years after randomization
Hemorrhagic stroke events | Within 3 years after randomization
Myocardial infarction events | Within 3 years after randomization
Proportion of patients achieving modified Rankin Scale score (mRS) 0-1 | At 3 years after randomization
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death], with higher scores indicating greater disability)
The score of mini-Montreal Cognitive Assessment | At 3 years after randomization
  The score of mini-Montreal Cognitive Assessment (range, 0 to 15, with higher scores indicating greater cognition)
Quality of life assessed by EuroQol 5 Dimensions 5 level questionnaire (EQ-5D-5L) | At 3 years after randomization
  The EQ-5D-5L includes 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= n
Rate of Falls | Within 3 years after randomization
All-cause death | Within 3 years after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The study is proceeding.